CLINICAL TRIAL: NCT04387526
Title: Efficacy and Safety of Sofosbuvir Plus Daclatasvir With or Without Ribavirin: Large Real-life Results of Patients With Chronic Hepatitis C Genotype 4
Brief Title: Sofosbuvir Plus Daclatasvir With or Without Ribavirin and Chronic HCV Genotype (GT) 4
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel-Gabbar, Ph.D, Associate Prof, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOF-DCV-RBV
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: Sofosbuvir; Daclatasvir; Ribavirin; HCV GT 4
MeSH Terms: interventions — daclatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SOF/DCV (Active Comparator): Easy to treat arm: Participants were treated with a dual therapy (SOF and DCV) for 12 weeks.
  This arm included non-cirrhotic treatment-naïve patients
  Interventions: Drug: (SOF and DCV)
- SOF/DCV/RBV + Cirrhosis (Active Comparator): This difficult-to-treat arm included 111 cirrhotic participants who were treated with a triple therapy (SOF, DCV, and RBV) for 12 weeks.
  Interventions: Drug: (SOF, DCV, and RBV)
- SOF/DCV/RBV + Non-Cirrhosis (Active Comparator): This difficult-to-treat arm included treatment-experienced non-cirrhotic participants (77 participants) who were treated with a triple therapy (SOF, DCV, and RBV) for 12 weeks.
  Interventions: Drug: (SOF, DCV, and RBV)

INTERVENTIONS:
Drug: (SOF and DCV)
  Other Names: Daklinza is a trade name of daclatasvir; Sovaldi is a trade name of sofosbuvir
  Arms: SOF/DCV
Drug: (SOF, DCV, and RBV)
  Other Names: Daklinza is a trade name of daclatasvir; Sovaldi is a trade name of sofosbuvir
  Arms: SOF/DCV/RBV + Cirrhosis; SOF/DCV/RBV + Non-Cirrhosis

SUMMARY:
This study aims to evaluate the efficacy and safety of DCV plus sofosbuvir (SOF) with or without ribavirin (RBV) for treatment of Egyptian participants infected with HCV GT4.

DETAILED DESCRIPTION:
Egyptian participants infected with HCV GT4 were classified into two groups: group 1 (easy to treat) was treated with a dual therapy of SOF/DCV daily for 12 weeks and group 2 (difficult to treat) was treated with a triple therapy of SOF/DCV/RBV daily for 12 weeks.

SOF dose was 400 mg/day given orally DCV was given in a dose of 60 mg/day, orally. RBV was given as oral tablets in the morning and in the evening based on patient's weight and tolerability (starting dose 600 mg/day to reach 1200 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Non-cirrhotic treatment-naïve participants
* FIB-4 < 3.25
* albumin > 3.5
* total bilirubin < 1.2 mg/dl
* international normalized ratio (INR) < 1.2
* platelet count > 150,000 mm3.
* experienced participants who had previously failed treatment with peg-IFN-α-/RBV, SOF/peg-IFN-α +RBV, or SOF/SMV
* Naïve cirrhotic participants were confirmed by ultrasonographic features of cirrhosis

Exclusion Criteria:

* liver disease of non-HCV etiology
* hepatitis B or human immune-deficiency virus (HIV) infection
* poorly controlled diabetic (HbA1C > 9) participants
* hepatocellular carcinoma
* a history of extra-hepatic malignancy within 5 years prior to the study
* pregnant or breast feeding
* renal disease; serum creatinine > 2.5 mg/dl or eGFR < 30 ml/min
* evidence of hepatic decompensation; INR > 1.7, serum albumin < 2.8 g/dl, total bilirubin > 3 mg/dl
* blood picture abnormalities such as anemia (hemoglobin concentration of 10 g/dl or less) and thrombocytopenia (platelet count < 50,000 cells/mm3)
* major severe illnesses such as congestive heart failure and respiratory failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) in Each Treatment Arm SVR12 | 12 weeks after last dose
  SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level < 15 IU/m 12 weeks after the last dose of drugs.
Number of Participants With Adverse Events in Each Treatment Arm | up for 12 weeks after planned End of Treatment (EOT).
  An adverse event (AE) is defined as any untoward medical occurrence in a participant clinical investigation after administering a pharmaceutical drugs
  Serious adverse event (SAE) is an event that results in death, life-threatening, requires hospitalization, or significant disability/incapacity

SECONDARY OUTCOMES:
Percentage of Participants With Viral relapse | 12 weeks after last dose
  Viral relapse was HCV RNA level ≤ 15 IU/ml at EOT, but detectable HCV RNA level > 15 IU/ml 12 weeks after planned EOT.
Percentage of Participants With On-treatment Virologic Failure | up tp 24 weeks
  On-treatment virologic failure was defined as quantifiable HCV RNA throughout the entire treatment period with HCV RNA greater than 15 IU/ml

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Moneim A, Aboud A, Abdel-Gabaar M, Zanaty MI, Ramadan M. Efficacy and safety of sofosbuvir plus daclatasvir with or without ribavirin: large real-life results of patients with chronic hepatitis C genotype 4. Hepatol Int. 2018 Jul;12(4):348-355. doi: 10.1007/s12072-018-9868-8. Epub 2018 May 12. PMID 29754329
- See also: This link describes the efficacy and safety of DCV plus sofosbuvir (SOF) with or without ribavirin (RBV) for treatment of Egyptian patients infected with HCV GT4. — https://doi.org/10.1007/s12072-018-9868-8